CLINICAL TRIAL: NCT03391596
Title: CareACT - Internet-based Intervention for Enhancing the Psychological Well-being of Elderly Caregivers
Brief Title: Internet-based Intervention for Enhancing the Psychological Well-being of Elderly Caregivers
Acronym: CareACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Gerocenter Foundation for Research and Development (Other)
Responsible Party: Principal Investigator, Riku Nikander, PhD, professor, The Gerocenter Foundation for Research and Development
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3E/2016
Record Dates: First submitted 2017-12-12; First posted 2018-01-05 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Depressive Symptoms; Psychological Distress; Quality of Life
Keywords: Family caregivers; Depressive symptoms; Psychological wellbeing; Internet-based intervention; Acceptance and Commitment Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based ACT intervention (Experimental): Group "Internet-based ACT intervention" will receive a 12-week Internet-based, acceptance and commitment therapy intervention
  Interventions: Behavioral: Internet-based ACT intervention
- Standardized rehabilitation (Active Comparator): Group "Standardized rehabilitation" will receive a standardized rehabilitation program in the rehabilitation center
  Interventions: Behavioral: Standardized rehabilitation
- Support by caregiver associations (Other): Group "Support by voluntary caregiver associations" will receive support given by caregiver associations
  Interventions: Behavioral: Support by voluntary caregiver associations

INTERVENTIONS:
Behavioral: Internet-based ACT intervention — The Internet-based ACT intervention is a 12-week program based on the processes of Acceptance and Commitment Therapy.
  Arms: Internet-based ACT intervention
Behavioral: Standardized rehabilitation — Standardized institutional rehabilitation in a rehabilitation center
  Arms: Standardized rehabilitation
Behavioral: Support by voluntary caregiver associations — Support given by voluntary caregiver associations
  Arms: Support by caregiver associations

SUMMARY:
This study will examine whether an Internet-based Acceptance and Commitment Therapy (ACT) intervention is effective, firstly, on reducing depressive symptoms, and, secondly, on improving well-being of elderly family caregivers. In our study, we will compare 1) the experimental Internet-based ACT group to 2) standardized institutional rehabilitation carried out in rehabilitation centers and to 3) support provided by voluntary family caregiver associations

DETAILED DESCRIPTION:
It is well-known that stress, low quality of life and depression are relatively common problems among family caregivers. The proportion of elderly family caregivers is rapidly increasing which emphasizes the need for new support systems. Internet-delivered psychological interventions are one possible approach, offering benefits as they are more easily to achieve for family caregivers who often are home-bound with their relatives.

This study will examine whether an Internet-based Acceptance and Commitment Therapy intervention would be effective, firstly, on reducing depressive symptoms, and, secondly, on improving well-being of elderly family caregivers.The family caregivers' depressive symptoms, perceived burden, anxiety, quality of life, psychological flexibility, personality and physical performance will be studied by a quasi-experimental study design comparing three groups of family caregivers (Group 1, experimental: Internet-based ACT intervention; Group 2, active comparator: Standardized institutional rehabilitation in a rehabilitation center; Group 3, other: Support given by voluntary family caregiver associations). Data collection will be performed at three time points: pre, 4 months and post (10 months).

Secondly, we also aim to examine demographics and psychological variables that could predict change in depression and perceived burden over time (pre, 4 months and post (10 months). A further aim of the study is to examine potential mediators on the effect of the interventions including psychological flexibility and suppression of thoughts. Moreover, we aim to study user experiences and satisfaction of the Internet-based program, i.e., how the family caregivers experience and accept the web-based ACT intervention.

ELIGIBILITY:
Inclusion Criteria for all groups:

* family caregiver
* at least 60 years of age

Inclusion Criteria for the experimental and active comparator group - depressive symptoms and/or psychological distress

Exclusion Criteria for all groups:

* parallel psychological treatment
* severe mental disorder

Additional inclusion criteria for the experimental group:

- computer and Internet connection or willingness to use a tablet provided by the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Inventory (BDI-II): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The BDI-II contains 21 questions about depressive symptoms and their severity. The scale ranges from 0 to 63 and the items are summed (0 to 13 indicates no or very few depressive symptoms, 14 to 19 indicates mild depression, 20 to 28 moderate depression, and 29 to 63 severe depression).

SECONDARY OUTCOMES:
Carers of Older People in Europe (COPE): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  COPE is an assessment of carers' perceptions of their role as caregiver: negative impact, positive value and quality of support of caregiving in informal carers of older people. It was developed in collaboration with several European countries as a brief first-stage assessment tool to identify caregivers who may need supportive interventions of any kind.
WHO Quality of Life-BREF (WHOQOL-BREF): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Generalized Anxiety Disorder 7-item (GAD-7) scale: change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of the four most common anxiety disorders (Generalized Anxiety Disorder, Panic Disorder, Social Phobia and Post Traumatic Stress Disorder). GAD-7 has seven items, which measure severity of various signs of GAD according to reported response categories with assigned points (Not at all: 0 points; Several days: 1 point; More than half the days: 2 points; and Nearly every day: 3 points). Assessment is indicated by the total score (min 0, max 21). Higher GAD-7 scores correlate with disability and functional impairment. 5-9 points indicate moderate anxiety, 10-14 moderate and >15 severe anxiety.
Sense of Coherence (SOC-13): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The SOC-13 is derived from the original 29-item scale measuring different aspects of sense coherence. Responses are made on a 7-point scale.The SOC-13 scale has three components: Comprehensibility (items 2, 6, 8, 9, 11; min 5, max 35), Manageability (items 3, 5, 10, 13; min 4, max 28) and Meaningfulness (items 1, 4, 7, 12; min 4, max 28) with higher scores indicating better outcomes. This scale is rated on a 7-point likert scale, a total score can also be used and the coding for items 1, 2, 3, 7 and 10 should be reversed. The subscales are combined to compute a total score. SOC scores range from 13 to 91 with higher scores indicating a better outcome: more sense of coherence.
Acceptance and Action Questionnaire (AAQ-II): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The AAQ-II is a measure with seven questions to be answered on a scale of 1 (never true) to 7 (always true) participant's willingness to be in contact with negative private events, acceptance of these events, and whether they can live in accordance with their values. Summation of the scores results in a total mark ranging from 7 to 49, whereby a higher score indicates means a higher level of psychological flexibility, e.g. higher acceptance.
Experiential Avoidance in Caregiving Questionnaire (EACQ): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The EACQ is a scale measuring experiential avoidance in the caregiving context: 1. Active Avoidant Behaviors, 2) Intolerance of Negative Thoughts and Emotions Towards the Relative and 3) Apprehension Concerning Negative Internal Experiences Related to Caregiving. The questionnaire consists of 15 items rated on a 5-point Likert scale. Each statement can be answered by 1: not at all, 2: a little, 3: somewhat, 4: often and 5: a lot. Factor 1 is made up of 6 items that measure caregivers' behaviors for avoiding negative thoughts related to caregiving (min 5, max 25). Factor 2 include 4 items with content related to rigid verbal thinking about negative emotions/thoughts with regard to the care-recipient (min 4, max 20), the factor 3 composes of 5 items referring to reluctant attitudes towards negative thoughts regarding the relative (min 5, max 25). The subscales are summed to compute a total score. Higher values represent more avoidance, e.g. worse outcome.
White Bear Suppression Inventory (WBSI): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The WBSI is a 15-item questionnaire that is designed to measure thought suppression. Chronic thoughts suppression is related to obsessive thinking and negative affect associated with depression and anxiety. The scoring of the WBSI is based on a 5 point scale from Strongly disagree (1) to Strongly agree (5). The total score (range from 15 to 75) is obtained by summing up the responses that are provided by respondents. Higher scores on the WBSI indicate greater tendencies to suppress thoughts.
The 'Short Five' (S5): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The Short Five personality questionnaire is a 60-item questionnaire constructed for measuring 30 facets of the Five-Factor Model
Short Physical Performance Battery (SPPB): change from baseline to 4 months and 10 months | baseline, 4 months, post (10 months)
  The Short Physical Performance Battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests (Guralnik et al., 2000). It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.

OTHER OUTCOMES:
User experiences questionnaire (developed by the research group) | 4 months (only experimental group)
  The questionnaire developed by the research group includes 9 questions investigating experiences of the intervention as a whole and assessed its most beneficial aspects. The first five questions are using a scale from 1 to 10 with answer options such as 1 = very unsatisfied, 10 = very satisfied (question 1); 1 = not at all important, 10 = very important (question 2 and 4); 1 = very satisfied, 10 = not at all satisfied (question 3); 1 = has deteriorated,10 = has improved remarkably (question 5). Question 6 assesses the current well-being situation including 7 options. Question 7 assesses weekly time spent in the web program with 4 different options (less than 1 hour, between 1-2 hours, 2-3 hours and more than 3 hours). The 2 last questions are open-ended questions.
Closing interview (developed by the research group) questions | 4 months (only experimental group)
  The questionnaire includes 9 questions investigating caregiver experiences with the web-based program. 5 of the questions are open-ended questions, 3 questions are close-ended questions which can be answered with Yes or No. Examples for questions: Question 1: What kind of experience was it to participate in this program? Question 3:What have you learned from this program?. Question 4: Was the program easy to use? One question (Would you recommend the web-program to other family caregivers?) includes a scale from 1 (not at all) to 10 (very likely).

CONTACTS AND LOCATIONS:
Overall Officials: Riku Nikander, Professor, Study Director — Gerocenter Foundation for Research and Development
Locations (1):
- Gerocenter Foundation for Research and Development, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lappalainen P, Pakkala I, Nikander R. CareACT - internet-based intervention for enhancing the psychological well-being of elderly caregivers - a study protocol of a controlled trial. BMC Geriatr. 2019 Mar 5;19(1):72. doi: 10.1186/s12877-019-1071-9. PMID 30836951